CLINICAL TRIAL: NCT01778296
Title: Repair of Soft Tissue Defect of the Finger Using the Heterodigital Neurocutaneous Island Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBTS1301283; CHS1301-00146 (Other: Hebei Clinical Trail Committee)
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2012-05

CONDITIONS: Sensory Reconstruction of the Volar Aspect of the Finger; The Heterodigital Neurocutaneous Island Flap
Keywords: Dorsal branch of the digital nerve;; dorsal digital artery;; dorsal digital island flap;; neurocutaneous island flap.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical flap (Experimental): The neurocutaneous island flap is based on the dorsal branch of the digital nerve
  Interventions: Device: the neurocutaneous island flap

INTERVENTIONS:
Device: the neurocutaneous island flap — The neurocutaneous island flap of the dorsal branch of the digital nerve can be used for repair the defects of the proximal and middle phalanxes of adjacent fingers.
  Other Names: dorsal digital island flap

SUMMARY:
The dorsum of the finger is a reliable flap donor site in reconstructive hand surgery because of its similar quality to the original. The dorsal digital island flap can be used for repairing the defect of adjacent finger, but the limited length of the pedicle precludes its use for a more distal defect. The heterodigital neurocutaneous island flap of the dorsal branch of the digital nerve can be used as an alternative to resolve this problem.

DETAILED DESCRIPTION:
At final follow-up, we measured the sensibility of the flaps using the Semmes-Weinstein monofilament test and the static 2-point discrimination test. The test points were at the center of the radial or ulnar portion of the pulp. The donor site, i.e. radial- or ulnar-dorsal aspect of the middle phalanx of the donor digit, was also evaluated. Each area was tested 3 times with a Discriminator (Ali Med, Dedham, MA). We stopped at 4mm as a limit of 2PD and considered this normal.

ELIGIBILITY:
Inclusion Criteria:

* the soft tissue defects involving the middle phalanx, the proximal interphalangeal joint, or both;
* a defect greater than or equal to 2 cm in length;
* a patient between 15 and 60 years of age.

Exclusion Criteria:

* concomitant injuries to the dorsal skin of the middle phalanx of adjacent finger that precluded its use as donor site;
* injuries to the course of donor nerve branch;
* a defect less than 1.5 cm in length;
* a fingertip or pulp defect;
* a soft tissue defect of the thumb.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Chen C, Zhang X, Shao X, Gao S, Wang B, Liu D. Treatment of a combination of volar soft tissue and proper digital nerve defects using the dorsal digital nerve island flap. J Hand Surg Am. 2010 Oct;35(10):1655-1662.e3. doi: 10.1016/j.jhsa.2010.07.011. PMID 20888502
- [Derived] Wang B, Zhao Y, Lu A, Chen C. Ulnar nerve deep branch compression by a ganglion: a review of nine cases. Injury. 2014 Jul;45(7):1126-30. doi: 10.1016/j.injury.2014.03.017. Epub 2014 Apr 3. PMID 24774037
- [Derived] Chen C, Tang P, Zhang L. Reconstruction of a soft tissue defect in the finger using the heterodigital neurocutaneous island flap. Injury. 2013 Nov;44(11):1607-14. doi: 10.1016/j.injury.2013.06.025. Epub 2013 Jul 18. PMID 23871427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February of 2008 to March of 2011,12 patients with soft tissue defects in the middle phalanx or the proximal interphalangeal joint were included in the study.The type of location is medical clinic. These patients were treated with the neurocutaneous island flap.
Pre-assignment Details: No wash out, run-in or transition happened in our study.
Period: Overall Study
Arm/Group | Surgical Flap
Started | 12 (There were 12 patients included in the study in the initial stage.)
Completed | 12 (No patient was lost to follow-up.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The participants with a follow-up period ≥18 months were included for this Baseline Measure.
Arm/Group | Surgical Flap
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  China | 12
Tissue reconstruction with the neurocutaneous island flap [Number; unit: participants] — The patients treated with the he neurocutaneous island flap are included in the study
  participants | 12 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Discriminatory Sensation of the Flap
Description: Discriminatory sensation of the flap is evaluated with the Static 2-point Discrimination Test. The test determines the minimal distance at which a subject can sense the presence of two needles. The modified American Society for Surgery of the Hand guidelines were used to stratify Discriminator measurements (excellent <6 mm; good 6-10 mm; fair 11-15 mm; poor >15 mm. The test point is at the center of the flap. Each area was tested 3 times with a Discriminator (Ali Med, Dedham, MA). Two out of 3 correct answers were considered proof of perception before proceeding to another lower value. We stop at 4mm as a limit of 2PD and considered this normal. These assessments take place at a single time point at the final follow-up.
Time Frame: 18 months to 24 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Surgical Flap
Number analyzed (Participants) | 12
mm | 8.3 (1.6)

2. Secondary Outcome: Cold Intolerance
Description: We access the cold intolerance of the injured and donor fingers using the self-administered Cold Intolerance Severity Score questionnaire10 that is rated into mild, moderate, severe, and extreme (0-25, 26-50, 51-75 and 76-100).
Time Frame: 18 months to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One year
Description: The only Adverse Event assessed for this study was Partial distal flap necrosis.
Arm/Group | Surgical Flap
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
The samples of our study are small, and the results may change as our experience grows.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes